CLINICAL TRIAL: NCT01478256
Title: A Comparative Study in the Clinical and Microbial Efficacy of Topical Besifloxocin Ophthalmic Suspension 0.6% With Erythromycin Ophthalmic Ointment 0.5% BID for the Management of Acute Blepharitis
Brief Title: Comparative Study in the Efficacy of Topical Besifloxocin With Erythromycin for the Management of Acute Blepharitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: John, George, M.D. (Industry)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Principal Investigator, George John, M.D., Prinicipal Investigator, John, George, M.D.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAIRB-11-0007
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Results first posted 2013-11-20 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-11

CONDITIONS: Blepharitis
Keywords: blepharitis; topical erythromycin; topical besifloxocin
MeSH Terms: conditions — Blepharitis | interventions — Erythromycin; besifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Besifloxocin (Active Comparator): Use of topical besifloxocin to treat acute blepharitis
  Interventions: Drug: Besifloxocin
- Erythromycin (Active Comparator): Topical Erythromycin ointment for treatment of acute blepharitis
  Interventions: Drug: Erythromycin

INTERVENTIONS:
Drug: Erythromycin — Topical erythromycin ointment twice a day
  Arms: Erythromycin
Drug: Besifloxocin — Topical Besifloxocin twice a day
  Other Names: Besivance
  Arms: Besifloxocin

SUMMARY:
This study looks at the improvements in signs and symptoms in patients with inflammation of the lids, blepharitis, using two different FDA approved topical antibiotic agents, Besifloxocin and Erythromycin. It also evaluates the bacterial cultures in these patients for microbiologic evidence of improvement.

DETAILED DESCRIPTION:
This is a pilot project involving thirty patients with a specific form of inflammtion of the lids called anterior blepharitis. The patients are graded for their signs a symptoms and then randomized to receive either topical Besifloxocin or Erythromycin in addition to standard lid hygiene measures. All patients have cultures of their eyelids performed prior to initiating therapy and are followed for four weeks. The antibiotics are used for two weeks following which repeat cultures of the lids are obtained. The patients are followed for one additional week to ensure that there is no recurrence of their symptoms once the antibiotics are discontinued.

Only adult patients (age 18-100)and women who are not of child bearing potential are included in this study. Then patients have to have symptoms and signs of the disease, blepharitis. Patient who are on unstable antibiotic or steroid regimens and those who cannot discontinue contact lens use are not included in this study.

ELIGIBILITY:
Inclusion Criteria:Acute blepharitis, age 18-100, Signs and symptoms of blepharitis -

Exclusion Criteria: women of child bearing potential, eye surgery within three months of study, contact lens wear, use of topical or antibacterial agents in past two weeks, use of topical or oral steroids in past two weeks unless stable dosage

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- George John, M.D., Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Besifloxocin: Use of topical besifloxocin twice a day to treat acute blepharitis
- Erythromycin: Topical Erythromycin ointment twice a day for treatment of acute blepharitis
Period: Overall Study
Arm/Group | Besifloxocin | Erythromycin
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Besifloxocin | Erythromycin | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (10) | 50 (12) | 49 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 7 | 8 | 15
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Signs and Symptoms of Blepharitis
Description: Signs and symptoms of blepharitis were scored and determined before and after treatment with two different antibiotics
Time Frame: Four weeks
Measure: Number; unit: participants
Arm/Group | Besifloxocin | Erythromycin
Number analyzed (Participants) | 15 | 15
participants | 15 | 15

2. Secondary Outcome: Evaluate Improvement of Bacterial Cultures With Two Different Topical Antibiotics
Description: Compare improvement of microbial cultures (greater inhibition of bacterial growth) with the two antibiotics used to treat blepharitis
Time Frame: Three weeks
Measure: Number; unit: participants
Arm/Group | Besifloxocin | Erythromycin
Number analyzed (Participants) | 15 | 15
participants | 15 | 15

ADVERSE EVENTS:
Arm/Group | Besifloxocin | Erythromycin
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No